CLINICAL TRIAL: NCT04006353
Title: A Phase 4, Single-center, Open-label, Parallel Study to Evaluate the Drug Interaction Between Albuvirtide (ABT) and Rifampin（RIF） in Healthy Adult Subjects
Brief Title: The Drug Interaction Between Albuvirtide (ABT) and Rifampin（RIF） in Healthy Adult Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Hongzhou Lu, professor, Shanghai Public Health Clinical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FB-ABWT-401
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Drug Interaction
MeSH Terms: interventions — albuvirtide; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: ABT (Experimental): Intravenous infusion of 320 mg ABT on Day 1, 2, 3, and 8.
  Interventions: Drug: ABT
- Group 2: ABT+RIF (Experimental): 600mg Rifampicin once daily from Day 1 to 16. Intravenous infusion of 320 mg ABT on Day 7, 8, 9 and 14.
  Interventions: Drug: ABT; Drug: RIF

INTERVENTIONS:
Drug: ABT — 320 mg, Intravenous infusion
  Other Names: albuvirtide
Drug: RIF — 600mg q.d.
  Other Names: rifampicin
  Arms: Group 2: ABT+RIF

SUMMARY:
This study is designed to estimate the drug interaction between RIF and ABT. This will be a single-center, open-label, parallel study in healthy adult subjects.

DETAILED DESCRIPTION:
The purpose of this study is to describe and compare RIF and ABT pharmacokinetics following administration of 320mg ABT and 600mg RIF.12 subjects will receive 320mg ABT on Days 1、2、3、8 (Treatment 1). And 12 subjects will receive 600mg RIF daily for 16 days from Day 1 to 16, and receive 320mg ABT on Days 7、8、9 and 14 (Treatment 2).

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age between 18 and 65 years；
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including physical examination, laboratory tests, Chest X-ray, abdominal B-ultrasound and ECG; No serious liver and kidney dysfunction, normal albumin value, and other indicators are in the normal range；
* Subjects weighing ≥50 kg and their BMI within the range 18.5-27.0 kg/m^2 (inclusive)；
* Agrees not to consume alcohol during the study；
* Both male and female subjects and their partners of childbearing potential agree to use contraception during the study；
* Females of childbearing potential must have a negative serum pregnancy test at Screening visit prior to receiving the first dose of study drug；
* ALT、AST、ALP and TBIL≤1×ULN；
* Willing and able to participate in all aspects of the study, including use of intravenous medication, completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent.

Exclusion Criteria:

* A positive anti-HIV-1 antibody result；
* A positive pre-study Hepatitis B surface antigen result；
* A Positive Hepatitis C antibody result；
* Syphilis infection as manifest by positive RPR；
* History of tuberculosis (TB) or lung disease；
* Currently active severe chronic diseases, metabolic diseases (such as diabetes), cardiovascular diseases, neurological and psychiatric diseases；
* Any known allergy or antibodies to the study drug or rifampicin；
* Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study；
* Active alcohol or drug abuse；
* Participation in an experimental drug trial(s) within 30 days or 5 half-lives of the Screening Visit；
* Currently active or chronic gastrointestinal dysfunction, or liver and kidney function disorders, would affect the absorption, metabolism, and/or excretion of the study drug. Subjects with a history of cholecystectomy, pepticulcer, inflammatory bowel disease or pancreatitis should be excluded；
* Use other prescription or over-the-counter medications, including vitamins, herbal medicines, or dietary supplements, 7 days prior to dosing or 5 half-life, unless the investigator believes that the drug will not interfere with the study procedure or compromise the safety of the subject；
* Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of ABT following ABT 320mg administration with and without RIF 600mg qd | Up to 17 days
  Pharmacokinetic(PK) parameters
Peak Plasma Concentration (Cmax) of RIF 600mg qd administration with and without ABT 320mg | Up to 17 days
  PK parameters
Area under the plasma concentration versus time curve (AUC) of ABT following ABT 320mg administration with and without RIF 600mg qd | Up to 17 days
  PK parameters
Area under the plasma concentration versus time curve (AUC) of RIF 600mg qd administration with and without ABT 320mg | Up to 17 days
  PK parameters

SECONDARY OUTCOMES:
Number of subjects with abnormal findings for laboratory parameters | Up to 17 days
  Number of subjects with Grade 3/4 laboratory parameters
Number of subjects with adverse events. | Up to 17 days
  An adverse event is any untoward medical occurrence in a clinical study subject, temporally associated with the use of a study treatment, whether or not considered related to the study treatment.
Number of subjects with severity of adverse events | Up to 17 days
  The Division of AIDS table for grading the severity of adult and pediatric adverse events will be used to assess severity.

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, Ph.D, Study Director — Shanghai Public Health Clinical Center
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No